CLINICAL TRIAL: NCT03764163
Title: Image and Model Based Analysis of Lung Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eric A. Hoffman (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Eric A. Hoffman, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 199708651; 5R01HL064368 (NIH)
Record Dates: First submitted 2018-03-30; First posted 2018-12-04 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Function Tests; Tomography, X-Ray Computed; Surveys and Questionnaires; Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Participants (Experimental): Pulmonary Function Test, Questionnaires, CT scans, perfusion scan, ventilation scan, Xenon gas ventilation CT scan with hyperpolarized 3-Helium MRI Scan.
  Interventions: Diagnostic Test: Pulmonary Function Test; Diagnostic Test: CT Scans; Behavioral: Questionnaires; Diagnostic Test: MRI; Biological: Xenon gas

INTERVENTIONS:
Diagnostic Test: Pulmonary Function Test — Spirometry, Diffusing Capacity of the Lungs (DLCO), Lung Volumes
Diagnostic Test: CT Scans — volume scans, perfusion scan, ventilation scan
Behavioral: Questionnaires — Human Subjects Questionnaire, Baseline Dyspnea Index, Chronic Respiratory Questionnaire
Diagnostic Test: MRI — proton scans, hyperpolarized 3-Helium scan
Biological: Xenon gas — ventilation CT scans

SUMMARY:
The purpose of this research study is to develop CT scanning and image analysis techniques to help define and measure several key properties of the pulmonary system that cannot be obtained by other tests or exams.

DETAILED DESCRIPTION:
Specifically, the investigators are interested in understanding the difference between the normal aging process and the events that lead to emphysema. Additionally, the investigators are interested in understanding the earliest signs (lung inflammation) of the disease process leading to three lung diseases, which include emphysema, fibrosis and sarcoidosis; all of which are described as "inflammatory lung diseases." The investigators will be using the data from this study to help define the normal values for the measured properties as well as deviation from normal values in smokers without defined lung disease and patients with inflammatory lung disease. The investigators believe that the analysis and scanning techniques being developed as part of this research will provide new and previously unavailable information on normal and diseased lungs so that ultimately the investigators can detect specific changes in the lungs due to a disease and measure any improvements in the anatomy and/or function of the pulmonary system after a patient has undergone treatment. This study involves research using X-Ray computed tomography (CT) scanner, which is similar to previous CT scanners but operates much faster and provides finer image detail.

ELIGIBILITY:
Inclusion Criteria:

* Non smokers, age 20-29, 40-49, 60-69, 80-89, cannot have smoked more than 20 cigarettes in their lifetime
* Smokers, age 20-29, 40-49, 60-69, 80-89, currently smoking a minimum of 1 pack (20 cigarettes) per day, normal smokers and mild to moderate Chronic Obstructive Pulmonary Disease (COPD)

Exclusion Criteria:

* Allergies - no allergies to shellfish, eggs, iodine
* Medications - no medications (except for birth control) for in the 'normal' category
* No asthma - as self reported
* BMI (Body Mass Index) - must not exceed 32 or 100kg of weight
* No other radiology studies in the last 12 months
* No metal in lung field - no metal from larynx to stomach
* No known heart disease
* No known kidney disease or diabetes
* Must not be pregnant - subjects of childbearing potential with be given a urine pregnancy test

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 1997-09-30 (Actual); Primary Completion 2015-06-05 (Actual); Study Completion 2015-06-05 (Actual)

PRIMARY OUTCOMES:
Normal lung aging assessed by CT imaging | up to 10 years
  Normal aging process of the lungs compared to common smoking related lung diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Hoffman, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
CT images will be shared including non-contrast images at TLC, FRC and RV as well as dual energy CT image data used to assess regional perfused blood volume. All associated pulmonary function test results will be shared. CT-derived metrics
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available starting 6 months after publication of the primary results of each aim
Access Criteria: Data will be provided to academic-based researchers upon written request to the PI, Eric A. Hoffman, PhD. A nominal charge will be made for the time it takes for a technician to prepare and transfer the requested data. This costs will not exceed $250. This service will be available for a minimum of 2 years of study close.